CLINICAL TRIAL: NCT04890444
Title: China Adrenal Disease Registry Study
Brief Title: China Adrenal Disease Registry
Acronym: CASE
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, Director, Head of Endocrinology, Principal Investigator, Clinical Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Ruijin-adrenal01
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Cushing Syndrome; Aldosteronism; Hypoadrenalism; Congenital Adrenal Hyperplasia; Adrenal Adenoma; Adrenal Incidentaloma; Adrenal Carcinoma; Pheochromocytoma
MeSH Terms: conditions — Cushing Syndrome; Hyperaldosteronism; Adrenal Insufficiency; Adrenal Hyperplasia, Congenital; ACTH Syndrome, Ectopic; Adrenal incidentaloma; Adrenal Cortex Neoplasms; Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiologic studies have revealed a tremendous increase in the prevalence of adrenal associated disease and related mortality worldwide. In order to meet all the therapeutic challenges in adrenal disease in China, CASE was founded in 2020. The objective of CASE is to launch an adrenal disease management model based on the Internet health information platform which allows the application and evaluation of adrenal disease treatment strategies at multiple centers. The proprietary electronic medical database will help the dynamic big-data analysis in epidemiology of adrenal disease, diagnosis, and treatment.

DETAILED DESCRIPTION:
In order to meet all the challenges in the diagnosis and treatment of adrenal diseases in China, CASE was founded in 2020. With advanced medical equipment and Internet of Things (IoT) technology, CASE is committed to creating an online and offline integrated solution for adrenal disease, and for the entire spectrum of adrenal disease, to achieve a more convenient and precise model of care for patients, aiming to establish a platform with diagnosis and treatment of adrenal disease and their long-term follow-up. It allows the application and evaluation of treatment strategies at these centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years old and ≤ 75 years
2. Patients diagnosed with adrenal associated diseases, including cushing syndrome, primary aldosteronism, primary hypoadrenalism, congenital adrenal hyperplasia and adrenal adenomas, incidentalomas, and carcinomas, pheochromocytoma, etc.
3. Provide written informed consent
4. Satisfactory compliance

Exclusion Criteria:

1. Patients with significantly reduced life expectancy (less than 2 years)
2. With Drug abuse
3. With AIDS or syphilis or infectious diseases such as viral tuberculosis in active phase at enrollment

Ages: 16 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational study. Participants enrolled in the study were diagnosed with adrenal associated diseases, including cushing syndrome, primary aldosteronism, primary hypoadrenalism, congenital adrenal hyperplasia and adrenal adenomas, incidentalomas, and carcinomas, pheochromocytoma. No gender restriction, between 16 and 75 years old.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of adrenal diseases in China | through study completion, an average of 1 year
Number of participants with complication of adrenal diseases in China | through study completion, an average of 1 year

SECONDARY OUTCOMES:
concentration of aldosterone | through study completion, an average of 1 year
concentration of cortisol | through study completion, an average of 1 year
concentration of urine cortisol | through study completion, an average of 1 year
concentration of androstenedione | through study completion, an average of 1 year
concentration of adrenocorticotropic hormone | through study completion, an average of 1 year
concentration of 17-hydroxyprogesterone | through study completion, an average of 1 year
concentration of metanephrines | through study completion, an average of 1 year
changes in adrenal CT | through study completion, an average of 1 year
percentage of hypoadrenalism | through study completion, an average of 1 year
Mental health status | through study completion, an average of 1 year
  The symptom checklist-90 will be used to evaluate the changes of participants' psychological state through study completion from 10 aspects, including somatization, obsessive-compulsive symptoms, interpersonal sensitivity, depression, anxiety, hostility, terror, paranoia, psychotic and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology, Shanghai, China

IPD SHARING:
Plan to Share IPD: No